CLINICAL TRIAL: NCT05226247
Title: Evaluation of the Role of Systolic Dysfunction in Weaning Failure Related to Weaning-induced Pulmonary Edema: the SystoWean Study
Brief Title: Systolic Function and Weaning-induced Pulmonary Edema (SystoWean Study)
Acronym: SystoWean
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-PP-28
Record Dates: First submitted 2022-01-18; First posted 2022-02-07 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Mechanical Ventilation Complication; Pulmonary Edema
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Intervention Model Description: Cohort Study
Masking Description: All echographic measurements will be analyzed offline, blinded to the patients' response to spontaneous breathing trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high-risk of weaning-induced pulmonary edema (Other): Critically-ill patients under mechanical ventilation for more than 48h, who are at high-risk of weaning-induced pulmonary edema and in whom the attending physician decided to perform a spontaneous breathing trial.
  Interventions: Procedure: Spontaneous breathing trial

INTERVENTIONS:
Procedure: Spontaneous breathing trial — To perform cardiac and lung echography before and during a spontaneous breathing trial

SUMMARY:
The purpose of this study is to determine if the left and right ventricular systolic function is involved in the development of weaning failure related to weaning-induced pulmonary edema.

DETAILED DESCRIPTION:
Weaning from mechanical ventilation remains a central step in the management of critically-ill patients, since weaning failure and prolonged duration of mechanical ventilation are not only associated with an increase in the length of stay in intensive care but also with greater morbidity and mortality. One of the well-recognized causes of weaning failure is weaning-induced pulmonary edema (WIPO), which accounts for almost 60% of the causes of weaning failure and ranging up to 75% in high-risk patients, i.e. patients with medical history of chronic heart disease, chronic respiratory failure and obesity.

Echocardiography is increasingly used in intensive care and allows non-invasive assessment of diastolic function as well as left ventricular (LV) and right (RV) systolic function, including during a spontaneous breathing test. Although LV diastolic dysfunction appears to be a major determinant of WIPO, the role of LV and RV systolic dysfunction is less unequivocal and has been poorly studied so far. Scarce data showed that patients experiencing WIPO tended to exhibit more frequently LV systolic dysfunction, as demonstrated by a lower LV ejection fraction (LVEF) and no study but two have investigated the potential role of RV systolic function. Moreover, assessing LV systolic function with LVEF measurement suffers from several limitations, especially in critically-ill patients.

Thus, the main goal of this study is to investigate whether LV and RV systolic function is involved in the development of WIPO. The second goal of this study is to determine the best echocardiographic parameter to assess LV and RV systolic function during the weaning process.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive mechanical ventilation for more than 48 hours
2. Patients indicated, according to intensivists, for carrying out a spontaneous breathing trial weaning test, based on the presence of all of the following criteria:

   1. SpO2> 90% with FiO2 ≤40% and PEEP ≤5 cmH2O
   2. Cough effectiveness on tracheal aspirations
   3. Lack of hemodynamic instability and of disorders of consciousness
3. Patients at high risk of weaning-induced pulmonary edema (WIPO), defined by one or more of the following criteria:

   1. Obesity, defined by a body mass index> 30 kg/m²
   2. Chronic obstructive pulmonary disease
   3. Chronic heart disease

Exclusion Criteria:

1. Age <18 years and pregnant women
2. Patients with a decision of not to resuscitate
3. Poor echogenicity
4. Severe mitral valve disease (leakage and/or stenosis, bioprosthesis)
5. Patients with pacemaker
6. Tracheostomy
7. Chronic neuromuscular or neurodegenerative diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing left and/or right ventricular | 24 months
  Left ventricular systolic function will be assessed by several

SECONDARY OUTCOMES:
Proportion of patients experiencing a weaning-induced pulmonary | 24 months
  WiPO is defined by new acute respiratory failure during spontaneous
Clinical and echocardiographic predictors of weaning-induced | 24 months
  To test the ability of different clinical and echocardiographic

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Dijon, Dijon
  - CHU de NICE, Nice
  - Hôpital Cochin, Paris

IPD SHARING:
Plan to Share IPD: No
No plan is established